CLINICAL TRIAL: NCT00274937
Title: Treatment of Childhood Nasopharyngeal Carcinoma With Neoadjuvant Chemotherapy and Concomitant Chemoradiotherapy: A Groupwide Phase III Study
Brief Title: Radiation Therapy, Amifostine, and Chemotherapy in Treating Young Patients With Newly Diagnosed Nasopharyngeal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARAR0331; NCI-2009-00412 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000454849; COG-ARAR0331; ARAR0331; ARAR0331 (Other: Children's Oncology Group); ARAR0331 (Other: CTEP); U10CA180886 (NIH); U10CA098543 (NIH)
Record Dates: First submitted 2006-01-10; First posted 2006-01-11 (Estimated); Results first posted 2017-01-19 (Estimated); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Stage I Nasopharyngeal Keratinizing Squamous Cell Carcinoma AJCC v7; Stage I Nasopharyngeal Undifferentiated Carcinoma AJCC v7; Stage II Nasopharyngeal Keratinizing Squamous Cell Carcinoma AJCC v7; Stage II Nasopharyngeal Undifferentiated Carcinoma AJCC v7; Stage III Nasopharyngeal Keratinizing Squamous Cell Carcinoma AJCC v7; Stage III Nasopharyngeal Undifferentiated Carcinoma AJCC v7; Stage IV Nasopharyngeal Keratinizing Squamous Cell Carcinoma AJCC v7; Stage IV Nasopharyngeal Undifferentiated Carcinoma AJCC v7
MeSH Terms: interventions — Amifostine; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Fluorouracil; dehydroftorafur; Radiotherapy; Radiation

ARMS (2):
- Stratum I (radiotherapy, chemoprotective agent) (Experimental): Patients undergo radiotherapy 5 days a week for 8 weeks. Patients also receive amifostine subcutaneously on the same days they undergo radiotherapy.
  Interventions: Drug: Amifostine; Other: Laboratory Biomarker Analysis; Radiation: Radiation Therapy
- Stratum II (chemotherapy, chemoprotective agent, radiotherapy) (Experimental): Patients receive cisplatin IV over 6 hours on day 1 and fluorouracil IV continuously on days 1-4. Treatment repeats every 3 weeks for 3 courses. In weeks 10-18, patients undergo radiotherapy and receive amifostine as in stratum I. Patients also receive 3 courses of cisplatin as before.
  Interventions: Drug: Amifostine; Drug: Cisplatin; Drug: Fluorouracil; Other: Laboratory Biomarker Analysis; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Amifostine — Given subcutaneously
  Other Names: Amifostine Trihydrate; Aminopropylaminoethylthiophosphoric Acid Trihydrate; APAETP; Cytofos; Ethiofos; Ethyol; Gammaphos; WR 2721; WR-2721; WR2721; YM-08310
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
  Arms: Stratum II (chemotherapy, chemoprotective agent, radiotherapy)
Drug: Fluorouracil — Given IV
  Other Names: 5 Fluorouracil; 5 Fluorouracilum; 5 FU; 5-Fluoro-2,4(1H, 3H)-pyrimidinedione; 5-Fluorouracil; 5-Fluracil; 5-Fu; 5FU; AccuSite; Carac; Fluoro Uracil; Fluouracil; Flurablastin; Fluracedyl; Fluracil; Fluril; Fluroblastin; Ribofluor; Ro 2-9757; Ro-2-9757
  Arms: Stratum II (chemotherapy, chemoprotective agent, radiotherapy)
Other: Laboratory Biomarker Analysis — Correlative studies
Radiation: Radiation Therapy — Undergo radiotherapy
  Other Names: Cancer Radiotherapy; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation

SUMMARY:
This phase III trial is studying how well radiation therapy, amifostine, and chemotherapy work in treating young patients with newly diagnosed nasopharyngeal cancer. Radiation therapy uses high-energy x-rays to kill tumor cells. Drugs, such as amifostine, may protect normal cells from the side effects of radiation therapy. Drugs used in chemotherapy, such as cisplatin and fluorouracil, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving radiation therapy together with amifostine and chemotherapy may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the response rate, overall survival, and event-free survival of children with advanced nasopharyngeal carcinoma who are treated with induction chemotherapy followed by concurrent chemoradiotherapy and amifostine.

SECONDARY OBJECTIVES:

I. Characterize the role of Epstein-Barr virus (EBV) in the pathogenesis of nasopharyngeal carcinoma in children.

II. Investigate the predictive value of the detection of EBV DNA in the peripheral blood of children with nasopharyngeal carcinoma.

III. Determine the incidence of NUT rearrangements in childhood nasopharyngeal carcinoma.

IV. Determine the radioprotective effect of amifostine when given daily prior to radiation therapy.

OUTLINE: This is a nonrandomized, multicenter study. Patients are stratified according to stage of disease (I or IIA [stratum I] vs IIB-IV [stratum II]).

STRATUM I: Patients undergo radiotherapy 5 days a week for 8 weeks. Patients also receive amifostine subcutaneously on the same days they undergo radiotherapy.

STRATUM II:

INDUCTION THERAPY (weeks 1-9): Patients receive cisplatin IV over 6 hours on day 1 and fluorouracil IV continuously on days 1-4. Treatment repeats every 3 weeks for 3 courses in the absence of disease progression or unacceptable toxicity. Patients with responding or stable disease proceed to consolidation therapy.

CONSOLIDATION THERAPY (weeks 10-18): Patients undergo radiotherapy and receive amifostine as in stratum I. Patients also receive cisplatin IV over 6 hours on days 1 and 22 (2 courses).

After completion of study treatment, patients are followed periodically for 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of nasopharyngeal carcinoma WHO type II or III

  * Stage I-IV disease
  * Newly diagnosed disease
* Performance status

  * Patients ≤ 16 years of age: Lansky 60-100%
  * Patients > 16 years of age: Karnofsky 60-100%
* Creatinine clearance or radioisotope glomerular filtration rate ≥ 70 mL/min
* Creatinine based on age/gender as follows:

  * No greater than 0.4 mg/dL (for patients 1 month to < 6 months of age)
  * No greater than 0.5 mg/dL (for patients 6 months to < 1 year of age)
  * No greater than 0.6 mg/dL (for patients 1-2 years of age)
  * No greater than 0.8 mg/dL (for patients < 6 years of age)
  * No greater than 1.0mg/dL (for patients 6 to < 10 years of age)
  * No greater than 1.2 mg/dL (for patients 10 to < 13 years of age)
  * No greater than 1.4 mg/dL (for female patients 13 to ≥ 16 years of age)
  * No greater than 1.5 mg/dL (for male patients 13 to < 16 years of age)
  * No greater than 1.7 mg/dL (for male patients ≥ 16 years of age)
* Bilirubin ≤ 1.5 times upper limit of normal (ULN) for age
* AST or ALT < 2.5 times ULN for age
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No prior chemotherapy or radiotherapy to the nasopharynx or neck for the treatment of nasopharyngeal carcinoma

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 111 (Actual)
Dates: Start 2006-02-20 (Actual); Primary Completion 2014-12-31 (Actual); Study Completion 2022-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Rodriguez-Galindo, Principal Investigator — Children's Oncology Group
Locations (109):
- United States (101):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kaiser Permanente Downey Medical Center, Downey, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Mattel Children's Hospital UCLA, Los Angeles, California
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - University of Connecticut, Farmington, Connecticut
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Lee Memorial Health System, Fort Myers, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Saint Mary's Hospital, West Palm Beach, Florida
  - Children's Healthcare of Atlanta - Egleston, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Riley Hospital for Children, Indianapolis, Indiana
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Helen DeVos Children's Hospital at Spectrum Health, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Nevada Cancer Research Foundation NCORP, Las Vegas, Nevada
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - New York Medical College, Valhalla, New York
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - Mercy Children's Hospital, Toledo, Ohio
  - University of Toledo, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Saint Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Greenville Cancer Treatment Center, Greenville, South Carolina
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Princess Margaret Hospital for Children, Perth, Western Australia, Australia
- Canada (7):
  - Alberta Children's Hospital, Calgary, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - IWK Health Centre, Halifax, Nova Scotia
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
  - Centre Hospitalier Universitaire de Quebec, Québec

REFERENCES:
- [Derived] Jeha S, Pei D, Choi J, Cheng C, Sandlund JT, Coustan-Smith E, Campana D, Inaba H, Rubnitz JE, Ribeiro RC, Gruber TA, Raimondi SC, Khan RB, Yang JJ, Mullighan CG, Downing JR, Evans WE, Relling MV, Pui CH. Improved CNS Control of Childhood Acute Lymphoblastic Leukemia Without Cranial Irradiation: St Jude Total Therapy Study 16. J Clin Oncol. 2019 Dec 10;37(35):3377-3391. doi: 10.1200/JCO.19.01692. Epub 2019 Oct 28. PMID 31657981
- [Derived] Rodriguez-Galindo C, Krailo MD, Krasin MJ, Huang L, McCarville MB, Hicks J, Pashankar F, Pappo AS. Treatment of Childhood Nasopharyngeal Carcinoma With Induction Chemotherapy and Concurrent Chemoradiotherapy: Results of the Children's Oncology Group ARAR0331 Study. J Clin Oncol. 2019 Dec 10;37(35):3369-3376. doi: 10.1200/JCO.19.01276. Epub 2019 Sep 25. PMID 31553639
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive — https://nctn-data-archive.nci.nih.gov/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No patients were enrolled to Stratum 1.
Groups:
- Stratum II: AJCC Stage IIb - IV
Period: Overall Study
Arm/Group | Stratum II
Started | 111
Completed | 91
Not Completed | 20
Not completed — Physician Decision | 10
Not completed — Withdrawal by Subject | 6
Not completed — Progressive Disease | 4

BASELINE CHARACTERISTICS:
Arm/Group | Stratum II
Number analyzed (Participants) | 111
Age, Continuous [Mean (Standard Deviation); unit: Participants] | 13.8 (2.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 75
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13
  Not Hispanic or Latino | 95
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 52
  White | 43
  More than one race | 0
  Unknown or Not Reported | 9
Region of Enrollment [Number; unit: participants]
  Canada | 2
  United States | 107
  Australia | 1
  Saudi Arabia | 1

OUTCOME MEASURES:

1. Primary Outcome: Two Year Event-free Survival (EFS)
Description: The two-year event-free survival will be compared with a standard established from adult oncology data and the results of POG-9486. The two-year Kaplan-Meier estimate of event-free survival will be compared with 70% using a 1-sided test of size 0.05 using the asymptotic distribution of the complementary log-log distribution of the estimate.
Time Frame: Up to Two Year After Enrollment
Population: No patients were enrolled to Stratum 1.
Measure: Number (95% Confidence Interval); unit: Estimated probability
Arm/Group | Stratum II
Number analyzed (Participants) | 111
Estimated probability | 0.87 [0.79 to 0.92]

2. Secondary Outcome: Predictive Value of Epstein-Barr Virus (EBV) DNA as Measured by Quantitative Detection at Enrollment on EFS 2 Years After Treatment
Description: Presence of EBV DNA in serum.
Time Frame: At study enrollment
Population: Data was and never will be collected.
Arm/Group | Stratum II
Number analyzed (Participants) | 0

3. Secondary Outcome: Prognostic Significance of EBV Viral Load
Description: Viral load in blood.
Time Frame: At study enrollment
Population: Data was and never will be collected.
Arm/Group | Stratum II
Number analyzed (Participants) | 0

4. Secondary Outcome: Predictive Value of the Detection of EBV DNA in the Peripheral Blood
Description: The prognostic value of the presence of EBV DNA will be assessed using the log-rank test, adjusted by initial stage of disease, if appropriate. The proposed analysis will take place at the analytic endpoint of the clinical trial.
Time Frame: Up to 6 years
Population: Funding was not obtained and results will never be reported.
Arm/Group | Stratum II
Number analyzed (Participants) | 0

5. Secondary Outcome: Protective Effects of Amifostine Assessed Primarily by Sialometry
Description: Weight of stimulated saliva production in grams.
Time Frame: At study enrollment
Population: Twenty-six patients in stratum 2 were evaluated at both study enrollment and at the end of consolidation for the weight of stimulated saliva production. This outcome measure was only collected for patients in Stratum 2.
Measure: Mean (Standard Deviation); unit: Grams of saliva
Arm/Group | Stratum II
Number analyzed (Participants) | 26
Grams of saliva
  At study Enrollment | 4.97 (5.44)
  At end of consolidation | 3.39 (4.71)

6. Secondary Outcome: Protective Effects of Amifostine Assessed Primarily by Sialometry: Weight of Unstimulated Saliva Production in Grams.
Description: Weight of unstimulated saliva production in grams.
Time Frame: At study enrollment
Population: Twenty-nine patients in stratum 2 were evaluated at both study enrollment and at the end of consolidation for the weight of unstimulated saliva production. This outcome measure was only collected for patients in Stratum 2.
Measure: Mean (Standard Deviation); unit: Grams of saliva
Arm/Group | Stratum II
Number analyzed (Participants) | 29
Grams of saliva
  At study Enrollment | 3.37 (4.49)
  At end of consolidation | 2.30 (3.90)

ADVERSE EVENTS:
Groups:
- Stratum II (Chemotherapy, Chemoprotective Agent, Radiotherapy): Patients receive cisplatin IV over 6 hours on day 1 and fluorouracil IV continuously on days 1-4. Treatment repeats every 3 weeks for 3 courses. In weeks 10-18, patients undergo radiation therapy and receive amifostine trihydrate as in stratum I. Patients also receive 3 courses of cisplatin as before.
  amifostine trihydrate: Given subcutaneously
  fluorouracil: Given IV
  cisplatin: Given IV
  laboratory biomarker analysis: Correlative studies
  radiation therapy: Undergo radiotherapy
Arm/Group | Stratum II (Chemotherapy, Chemoprotective Agent, Radiotherapy)
Serious Adverse Events (participants affected / at risk) | 79/111
Other Adverse Events (participants affected / at risk) | 36/111
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stratum II (Chemotherapy, Chemoprotective Agent, Radiotherapy) (N=111)
Abdominal infection (Infections and infestations) | 3
Abdominal pain (Gastrointestinal disorders) | 2
Acidosis (Metabolism and nutrition disorders) | 1
Activated partial thromboplastin time prolonged (Investigations) | 1
Acute kidney injury (Renal and urinary disorders) | 4
Alanine aminotransferase increased (Investigations) | 2
Allergic reaction (Immune system disorders) | 1
Anemia (Blood and lymphatic system disorders) | 9
Anorexia (Metabolism and nutrition disorders) | 19
Anxiety (Psychiatric disorders) | 1
Apnea (Respiratory, thoracic and mediastinal disorders) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 2
Cardiac troponin I increased (Investigations) | 1
Catheter related infection (Infections and infestations) | 2
Cheilitis (Gastrointestinal disorders) | 1
Chronic kidney disease (Renal and urinary disorders) | 2
Constipation (Gastrointestinal disorders) | 4
Dehydration (Metabolism and nutrition disorders) | 15
Depression (Psychiatric disorders) | 1
Dermatitis radiation (Injury, poisoning and procedural complications) | 1
Dry mouth (Gastrointestinal disorders) | 7
Dysphagia (Gastrointestinal disorders) | 11
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 1
Edema face (General disorders) | 1
Ejection fraction decreased (Investigations) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 2
Esophageal pain (Gastrointestinal disorders) | 2
Esophagitis (Gastrointestinal disorders) | 4
Eye infection (Infections and infestations) | 1
Fatigue (General disorders) | 5
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Fever (General disorders) | 1
Gastritis (Gastrointestinal disorders) | 2
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 2
Hearing impaired (Ear and labyrinth disorders) | 18
Heart failure (Cardiac disorders) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 9
Hyperkalemia (Metabolism and nutrition disorders) | 5
Hypermagnesemia (Metabolism and nutrition disorders) | 1
Hyperuricemia (Metabolism and nutrition disorders) | 2
Hypocalcemia (Metabolism and nutrition disorders) | 7
Hypokalemia (Metabolism and nutrition disorders) | 14
Hypomagnesemia (Metabolism and nutrition disorders) | 9
Hyponatremia (Metabolism and nutrition disorders) | 10
Hypophosphatemia (Metabolism and nutrition disorders) | 10
Hypotension (Vascular disorders) | 3
Infections and infestations - Other, specify (Infections and infestations) | 5
Investigations - Other, specify (Investigations) | 1
Laryngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1
Lip infection (Infections and infestations) | 1
Lymphocyte count decreased (Investigations) | 12
Mucositis oral (Gastrointestinal disorders) | 27
Nausea (Gastrointestinal disorders) | 25
Neck pain (Musculoskeletal and connective tissue disorders) | 2
Neutrophil count decreased (Investigations) | 27
Non-cardiac chest pain (General disorders) | 1
Oral pain (Gastrointestinal disorders) | 9
Pain (General disorders) | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 1
Peripheral motor neuropathy (Nervous system disorders) | 1
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 5
Pharyngitis (Infections and infestations) | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 5
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1
Radiation recall reaction (dermatologic) (Injury, poisoning and procedural complications) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Restrictive cardiomyopathy (Cardiac disorders) | 1
Seizure (Nervous system disorders) | 3
Sepsis (Infections and infestations) | 1
Sinus tachycardia (Cardiac disorders) | 1
Sinusitis (Infections and infestations) | 1
Skin infection (Infections and infestations) | 1
Small intestine infection (Infections and infestations) | 1
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 2
Stomach pain (Gastrointestinal disorders) | 1
Syncope (Nervous system disorders) | 2
Trismus (Musculoskeletal and connective tissue disorders) | 2
Vaginal infection (Infections and infestations) | 1
Vascular access complication (Injury, poisoning and procedural complications) | 2
Ventricular fibrillation (Cardiac disorders) | 1
Ventricular tachycardia (Cardiac disorders) | 1
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 21
Weight loss (Investigations) | 8
White blood cell decreased (Investigations) | 20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stratum II (Chemotherapy, Chemoprotective Agent, Radiotherapy) (N=111)
Constipation (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Dizziness (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 1
Ear pain (Ear and labyrinth disorders) | 1
Esophageal pain (Gastrointestinal disorders) | 1
Fever (General disorders) | 3
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1
Headache (Nervous system disorders) | 1
Hearing impaired (Ear and labyrinth disorders) | 29
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Insomnia (Psychiatric disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Salivary duct inflammation (Gastrointestinal disorders) | 1
Sinus bradycardia (Cardiac disorders) | 1
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 2
Vomiting (Gastrointestinal disorders) | 3
Weight loss (Investigations) | 1
White blood cell decreased (Investigations) | 2

LIMITATIONS AND CAVEATS:
Data was and never will never be collected for Outcome Measure #2 and Outcome Measure #3. Funding was not obtained and results will never be reported for Outcome Measure #4.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain prior Sponsor approval.